CLINICAL TRIAL: NCT01018901
Title: Goals for Sexual Functioning of Prostate Cancer Survivors and Their Partners Following Cancer Treatment
Brief Title: Goals of Sexual Function in Prostate Cancer Survivors and Their Partners After Cancer Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UPCC 23808
Record Dates: First submitted 2009-11-23; First posted 2009-11-24 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (Experimental): Patients and their partners complete surveys. Sexual function of men is assessed by the International Index of Erectile Function; sexual function of women is assessed by the Female Sexual Function Index.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Patients complete survey

SUMMARY:
RATIONALE: Gathering information about survivors of prostate cancer and their partners may help doctors learn more about the goals for sexual functioning after cancer treatment. PURPOSE: This clinical trial is studying the goals of sexual functioning in prostate cancer survivors and their partners after cancer treatment.

DETAILED DESCRIPTION:
Detailed DescriptionOBJECTIVES:

I. To collect data on the goals of sexual functioning among prostate cancer survivors and their partners following cancer treatment in order to identify specific components of interventions for future grant submissions on the psychosexual needs of prostate cancer survivors.

OUTLINE:

Patients and their partners complete surveys. Sexual function of men is assessed by the International Index of Erectile Function; sexual function of women is assessed by the Female Sexual Function Index.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer survivors who are: willing and able to provide informed consent; able to read, write, and speak English; married or are in married-like relationship; completed radiation or surgery for their prostate cancer 6 months to 5 years ago
* Partners of prostate cancer survivors must be: willing and able to provide informed consent; able to read, write, and speak English

Exclusion Criteria:

* Prostate cancer survivors will be excluded if they have undergone androgen deprivation therapy within the past 6 months and if their partners refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Goals of sexual functioning | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James Coyne, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States